CLINICAL TRIAL: NCT05850325
Title: Novel Exercises to Facilitate Recovery of Supination and Pronation for Distal Radius Fractures Managed With a Volar Plate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Indiana Hand to Shoulder Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR VP ROM
Record Dates: First submitted 2023-04-18; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Elbow Flexed at 90 Degrees (Other): subjects will be instructed to exercise the forearm with the elbow positioned by their side, in 90° of flexion.
  Interventions: Other: Group 1 Elbow Flexed at 90 Degrees
- Group 2: Elbow Fully Flexed (Experimental): subjects will be instructed to exercise the forearm with their elbow fully flexed to achieve supination and the elbow extended to achieve pronation.
  Interventions: Other: Group 2 Elbow Fully Flexed

INTERVENTIONS:
Other: Group 1 Elbow Flexed at 90 Degrees — subjects will be instructed to exercise the forearm with the elbow positioned by their side, in 90° of flexion.
  Other Names: Elbow Flexed to 90 Degrees
  Arms: Group 1: Elbow Flexed at 90 Degrees
Other: Group 2 Elbow Fully Flexed — subjects will be instructed to exercise the forearm with their elbow fully flexed to achieve supination and the elbow extended to achieve pronation.
  Other Names: Elbow Fully Flexed
  Arms: Group 2: Elbow Fully Flexed

SUMMARY:
The primary objective of this study is to evaluate the influence of elbow position on achieving forearm supination and pronation and wrist ROM postoperatively. It is anticipated the results will show recovery of functional motion in a shorter period of time (27 days average). As for the secondary objective of the study, it is anticipated there will be limited pain and cost-containment. These data elements will serve as secondary factors to evaluate.

DETAILED DESCRIPTION:
The current standard of care for forearm range of motion exercises is to position the elbow in 90 degrees of flexion at the side of the body for both supination and pronation.5,6 This study will compare standard of care forearm rotation exercises to exercising with the elbow in extension to facilitate pronation and exercising with the elbow in full flexion to facilitate supination in patients who have undergone surgery with a volar plate for distal radius fractures. We hypothesize that forearm motion will be achieved in a shorter number of days and with a greater arc of motion when the exercises are done in extremes of elbow flexion and extension.

This will be a prospective, unblinded, randomized study to evaluate forearm range of motion across two groups:

Control Group: subjects will be instructed to exercise the forearm with the elbow positioned by their side, in 90° of flexion.

Test Group: subjects will be instructed to exercise the forearm with their elbow fully flexed to achieve supination and the elbow extended to achieve pronation.

Randomization will occur post-operatively after the patient has signed consent to participate. Randomization will occur through a computerized random allocation and groups will be assigned by the Clinical Research Manager or designee.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects 18 years of age and older

  * Subjects with distal radius fractures with a volar plate
  * Subjects attending therapy at the Indiana Hand to Shoulder Center or affiliated satellites.
  * Subjects that attend the initial therapy visit between 5 and 10 days postoperative and begin the home therapy program (patient handout)

Exclusion Criteria:

* • Subjects under the age of 18

  * Additional surgical procedures or other factors preventing early active ROM of the forearm and/or wrist within the initial 10 days following surgery
  * Pre-existing medical conditions or injuries with resultant limitation in elbow, forearm or wrist ROM, patient-reported limited function, or limited ability to comply with home program (cognitive skills).
  * While undergoing therapy the initial 6 weeks, subjects provided with custom-fabricated or pre-fabricated devices, orthoses, or braces for the specific purpose of passively improving ROM of the elbow, forearm or wrist during the initial 6 weeks of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 6 Months
  forearm supination and pronation and wrist ROm

SECONDARY OUTCOMES:
Upper Limb Functional Index (ULFI) | 6 Months
  PROM functional questionnaire
QuickDisability of the Arm Shoulder Hand (DASH) | 6 Months
  PROM - functional questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No